CLINICAL TRIAL: NCT04757441
Title: Effects of ELDOA on Hamstring Tightness in Individuals With Non-Specific Low Back Pain.
Brief Title: Effects of ELDOA on Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00763 Sana Rasool
Record Dates: First submitted 2021-02-02; First posted 2021-02-17 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Non-specific Low Back Pain
Keywords: ELDOA; LBP; ROM; Flexibility; ODI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Conventional Treatment + Elongation Longitudinaux Decoaption of Osteo-Articulaire (ELDOA) (Experimental): Participants will receive conventional treatment along with ELDOA stretching exercises protocol at L5, S1.
  Interventions: Other: Group A: Conventional Treatment + Elongation Longitudinaux Decoaption of Osteo-Articulaire
- Group B: Conventional treatment (Other): Participants will receive only conventional treatment (Control)
  Interventions: Other: Group B: Conventional treatment

INTERVENTIONS:
Other: Group A: Conventional Treatment + Elongation Longitudinaux Decoaption of Osteo-Articulaire — ELDOA position for L5, S1 level Patient will ask to lie on his back, wedge buttocks in the corner of wall and raise his legs. Then Stretch the legs and push the heels toward ceiling. Extend the spine and stretch the arms above head .
  • Patient will hold this position for one minute and repeat it for 4 -5 times.
  Conventional treatment will include:
  * Hot pack for 15 minutes .
  * TENS for 10 minutes .
  * self stretching of hamstrings
  Arms: Group A: Conventional Treatment + Elongation Longitudinaux Decoaption of Osteo-Articulaire (ELDOA)
Other: Group B: Conventional treatment — Participants will receive only conventional treatment which will include:
  * Hot pack for 15 minutes .
  * TENS for 10 minutes .
  * self stretching of hamstrings
  Arms: Group B: Conventional treatment

SUMMARY:
The purpose of this study is to find the effects of ELDOA in increasing hamstring length in patients with nonspecific low back pain.This research will bring awareness about the concept of ELDOA exercises among clinicians and people to understand its benefits for treating back pain issues. Further, it will provide an important addition to the evidence-based treatment intervention of ELDOA

DETAILED DESCRIPTION:
Low back pain is the most commonly reported musculoskeletal condition, associated with injury and disability in adults worldwide. It is the leading cause of activity limitation and work absence throughout much of the world . Over 70% to 80% people experience low back pain somewhat once in their lives . Low back pain affects people of all ages, from children to the elderly, but it is more prevalent in young adults. Low back pain can lead to decrease in lumbar range of motion, change in gait pattern, and change of rhythm in the pelvis, limitations that can restrict social activities. Approximately more than 85% low back pain cases are categorized as non specific low back pain. Non-specific low back pain is defined as low back pain not attributable to a recognizable, known specific pathology (e.g, infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome) Hamstrings muscle is a postural muscle and as it is biarticular, it has tendency to shorten even under normal circumstances . Hamstrings are more prone to adaptive shortening than all other muscles of body .prevalence and incidences of Hamstrings tightness in non-specific low back pain individuals is high due to limited activity and lack of regular exercise . The hamstrings length is an essential component in the basic movements of the human body like walking and running . It is composed of three separate muscles; include semitendinosus, semimembranosus and biceps femoris which are present in the posterior part of thigh and help in the flexion of knee and extension of hip joint . Due to the attachment of hamstring muscles to the ischial tuberosity, the tightness of the hamstring produces posterior pelvic tilt which stops the flexion of hips during forward bending so reducing the lordosis of the lumbar spine. It may impair spinal loading and alter the Lumbar Pelvic Rhythm which will generate more strain on the lumbar segment giving rise to low back pain.

ELDOA stands for elongation Longitudinaux avec Decoaption Osteo-Articulaire, or LOADS (Longitudinal Osteo-Articular Decoaption Stretching). A system of exercises and movements that uses the center of gravity and locates a target area of the spine that needs to be either mobilized or re-aligned by placing and maintaining tension on the fascia, was developed by Guy Voyer in Europe more than 30 years ago . The purpose of ELDOA is to help manage stress and create space in the vertebral joints, allowing muscles to move freely. The results of these stretches include joint mobility, increased absorption of fluid within the discs of the spine, flexibility, improved muscle tone, postural alignment, body-mind connection, and coordination. The tension and release created by these stretches help normalize the posture.

In March-June 2019, a quasi- experimental study of 34 participants was conducted on Elongation Longitudinaux Avec Decoaption Osteo-Articulaire (ELDOA) in Lumbar Disc Protrusion. Two randomized group of patients with lumbar disc protrusion were treated and concluded that ELDOA improved pain and functional status of patients .

In Jan-June 2019, another quasi-experimental study conducted with 20 patients, Elongation Longitudinaux Avec Decoaption Osteo-Articulaire (ELDOA) in Cervical Disc Protrusion. ELDOA technique was compared with conventional physical therapy treatment. The results showed, improved functional status and pain.

In May 2019, an article published in Dynamic Chiropractic, Cervical spine degeneration- Exam to ELDOA founded significant results on using ELDOA exercises as main treatment intervention for cervical spine degeneration.

In 2019, A study inquired the combination effect of core stability and contract relax exercise on hamstring flexibility and concluded that the combination of both core stability and contract relax exercise better than core stability exercises only and as good as contract relax exercises in increasing hamstring flexibility

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for at least 2 months.
* A passive SLR angle of 70° or less.
* Both genders.
* 25-40 years age.
* Pain > 3 on NPRS

Exclusion Criteria:

* Any fracture of spine or lower limb.
* No neurological signs.
* Malignancy, infection, trauma or any bony deformity.
* Surgery of spine or lower limb.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Sit and Reach Test | 12th day
  Used for measurement of flexibility of the lower back and hamstring muscles.The reliability with ICC= 0.99 Baseline,6th visit,12th visit
Straight Leg Raise Passive Knee Extension Test (PKE) | 12 Day
  Examine the joint range and its quality of movement; in particular, the 'end feel' of the joint.It has excellent test-retest reliability with ICC=0.94 and moderate validity= 0.57 to 0.63 Baseline,6th visit,12th visit
The Oswestry Disability Index (ODI) | 12 Day
  Tool used to assess disability related to pain in individuals with acute, sub-acute, or chronic LBP. The total score of ODI range from 0 (no disability) to 100 (maximum disability). The ODI score is recommended as a back pain-specific measure of disability. Reliability with ICC= 0.85 and validity=0.77 Baseline,6th visit,12th visit

SECONDARY OUTCOMES:
Numeric pain rating scale | 12th day
  A scale for pain measurement, ranging from '0' representing no pain to '10' representing the worst or severe pain. The reliability with ICC= 0.64 to 0.86 Baseline,6th visit,12th visit
Inclinometer | 12th day
  It is an instrument used to measure range of motion (ROM) (36). The inter rater reliability with ICC= 0.80 Baseline,6th visit,12th visit

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Baharam NS, Hisham MY, Mohan V, Mohamad N. EFFECT OF STATIC STRETCHING ON MUSCLE ACTIVATION DURING SIT TO STAND AMONG LOW BACK PAIN POPULATION. Jurnal Teknologi. 2016;78(6-8)
- [Background] Tafazzoli F, Lamontagne M. Mechanical behaviour of hamstring muscles in low-back pain patients and control subjects. Clin Biomech (Bristol). 1996 Jan;11(1):16-24. doi: 10.1016/0268-0033(95)00038-0. PMID 11415594
- [Background] Jandre Reis FJ, Macedo AR. Influence of Hamstring Tightness in Pelvic, Lumbar and Trunk Range of Motion in Low Back Pain and Asymptomatic Volunteers during Forward Bending. Asian Spine J. 2015 Aug;9(4):535-40. doi: 10.4184/asj.2015.9.4.535. Epub 2015 Jul 28. PMID 26240711
- [Background] Seif HE, Alenazi A, Hassan SM, Kachanathu SJ, Hafez AR. The Effect of Stretching Hamstring, Gastrocnemius, Iliopsoas and Back Muscles on Pain and Functional Activities in Patients with Chronic Low Back Pain: A Randomized Clinical Trial. Open Journal of Therapy and Rehabilitation. 2015;3(04):139.
- [Background] Burton AK, Balague F, Cardon G, Eriksen HR, Henrotin Y, Lahad A, Leclerc A, Muller G, van der Beek AJ; COST B13 Working Group on Guidelines for Prevention in Low Back Pain. Chapter 2. European guidelines for prevention in low back pain : November 2004. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S136-68. doi: 10.1007/s00586-006-1070-3. No abstract available. PMID 16550446
- [Background] Moon JH, Jung JH, Won YS, Cho HY. Immediate effects of Graston Technique on hamstring muscle extensibility and pain intensity in patients with nonspecific low back pain. J Phys Ther Sci. 2017 Feb;29(2):224-227. doi: 10.1589/jpts.29.224. Epub 2017 Feb 24. PMID 28265144
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Jonhagen S, Nemeth G, Eriksson E. Hamstring injuries in sprinters. The role of concentric and eccentric hamstring muscle strength and flexibility. Am J Sports Med. 1994 Mar-Apr;22(2):262-6. doi: 10.1177/036354659402200218. PMID 8198197
- [Background] Hertling D, Kessler RM. Management of common musculoskeletal disorders: physical therapy principles and methods: Lippincott Williams & Wilkins; 2006
- [Background] Na'ima AL, Sari GM, Utomo DN, editors. Combination effect of core stability exercise and contract relax exercise on hamstring flexibility. Journal of Physics: Conference Series; 2019: IOP Publishing.
- [Background] Worrell TW, Perrin DH, Gansneder BM, Gieck JH. Comparison of isokinetic strength and flexibility measures between hamstring injured and noninjured athletes. J Orthop Sports Phys Ther. 1991;13(3):118-25. doi: 10.2519/jospt.1991.13.3.118. PMID 18796850
- [Background] Yildirim MS, Ozyurek S, Tosun O, Uzer S, Gelecek N. Comparison of effects of static, proprioceptive neuromuscular facilitation and Mulligan stretching on hip flexion range of motion: a randomized controlled trial. Biol Sport. 2016 Mar;33(1):89-94. doi: 10.5604/20831862.1194126. Epub 2016 Feb 8. PMID 26929476